CLINICAL TRIAL: NCT02382172
Title: Social Cognition and Interaction Training for Autism (SCIT-A)
Brief Title: Social Cognition and Interaction Training for Autism
Acronym: SCIT-A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other); Carolina Institute for Developmental Disabilities (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 14-2804
Record Dates: First submitted 2015-02-23; First posted 2015-03-06 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Autism; Social Behavior
MeSH Terms: conditions — Autistic Disorder; Social Behavior | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Social Cognition and Interaction Training for Autism (SCIT-A) (Experimental): The measures the investigators are giving assess participants' initial level of social deficits and the extent to which the therapy did or did not help their social skills. The research team will compare the level of difficulty that participants first reported with their subjective evaluation of their experience in the group sessions to determine whether the program is clinically useful for further development. The investigators will also have the participants complete eye tracking paradigms to assess possible changes in social functioning after completing the Social Cognition and Interaction Training for Autism (SCIT-A) program.
  Interventions: Behavioral: Social Cognition and Interaction Training for Autism (SCIT-A)
- Treatment As Usual (TAU) (Other): Continuation of services being given upon study entry.
  Interventions: Other: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Social Cognition and Interaction Training for Autism (SCIT-A) — The group therapy program is aimed at improving social cognitions and skills of individuals who find social situations difficult, stressful and/or uncomfortable and with a desire to enhance skills required for social interactions.
  Arms: Social Cognition and Interaction Training for Autism (SCIT-A)
Other: Treatment as Usual (TAU) — Participants in the treatment as usual (TAU) group will continue to receive other interventions (e.g., individual therapy, job skills coaching) during the Social Skills Clinic. No participants in either group will participate in other group-based interventions concurrently with their participation in this study.
  Arms: Treatment As Usual (TAU)

SUMMARY:
Purpose: To collect outcome measures such as eye tracking and questionnaire data prior to and following a group based clinical therapy program to determine the effectiveness of the therapy approach. The therapy program is aimed at improving social cognitions and skills of individuals who find social situations difficult, stressful and/or uncomfortable and with a desire to enhance skills required for social interactions.

Participants: Cohorts of individuals aged 10-69 years old with symptoms of a neurodevelopment disorder, who have general difficulty with social interactions.

Procedures: Participants enrolled in a clinical therapy program for improvement of social cognitions and skills will complete eye tracking tasks, several questionnaires and rating scales, and a diagnostic interview prior to and following the 8 week therapy program. The post treatment assessments will be conducted within a week of the therapy completion and then again approximately 2 months after the last therapy session. The entire study duration is expected to be approximately 17 weeks. These outcome measures will measure the effectiveness of the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 13-69.
2. Symptoms of a neurodevelopmental disorder.
3. English as primary language and ability to speak in fluent, full length sentences: Treatment will be conducted in a group setting in English.

Exclusion Criteria:

1. Inability to speak English fluently.

Ages: 10 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-01; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change in visual attention from baseline as measured by the Tobii Eye Tracking Paradigm | The pre-treatment assessment will take place within a week of beginning the social skills group. Immediately after the 8-week clinic, there will be another assessment and then a final assessment 2 months following completion of the therapy.
  Participants will complete an eyetracking task both before and after the Social Skills training clinic. The eyetracking task will be presented on a Tobii 1750 eyetracker integrated with a 17" display monitor (Tobii Technology, Stockholm, Sweden). The task will be an interactive visual exploration task that is a validated measure of social attention. It's a 15-minute eye tracking task, which is non-invasive and completely safe. During the task, participants will be asked to look at two children playing together. The Tobii eyetracker will record where the participants focus their gaze and for how long.

SECONDARY OUTCOMES:
Change in patient social skills as measured by the Social Responsiveness Scale (SRS) | The pre-treatment assessment will take place within a week of beginning the social skills group. Immediately after the 8-week clinic, there will be another assessment and then a final assessment 2 months following completion of the therapy.
  Each item is rated on a scale from 0 (never true) to 3 (almost always true). The SRS total raw score ranges from 0 to 195; a higher score indicates greater severity of social impairment.
Change in patient social cognition as measured by the Hinting Task | The pre-treatment assessment will take place within a week of beginning the social skills group. Immediately after the 8-week clinic, there will be another assessment and then a final assessment 2 months following completion of the therapy.
  This is a measure of Theory of Mind (ToM, i.e. ability to understand others' mental states). It consists of ten short vignettes involving social interactions between two characters, one of whom drops a hint at the end of the vignette about their desire or intention. The participant is asked to infer what the character means by their hint. This task will be completed at all testing visits. All participant groups will be asked to complete the Hinting task.
Change in patient social cognition as measured by the Penn Emotion Recognition Task-40 (ER40) | The pre-treatment assessment will take place within a week of beginning the social skills group. Immediately after the 8-week clinic, there will be another assessment and then a final assessment 2 months following completion of the therapy.
  This task measures face processing and emotion perception. The ER40 is a standardized test of facial emotion recognition ability consisting of color photographs of evoked expressions from adult actors displaying four basic emotions (happy, sad, angry, and fearful) and neutral facial expressions. This task takes approximately 5 minutes to complete and will be administered at each testing visit. All participant groups will be asked to complete the ER40 task.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Dichter, MA, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Carolina Institute for Developmental Disabilities, Carrboro, North Carolina, United States